CLINICAL TRIAL: NCT06934161
Title: Comparison of the Effectiveness of Innovative Techniques to Prevent Tissue Overheating During Corticotomy Using Smartphone-Based Thermography: Reticulated Surgical Guide vs Dynamic Navigation. A Split-mouth Randomized Pilot Clinical Trial.
Brief Title: Comparison of the Effectiveness of Innovative Techniques to Prevent Tissue Overheating During Corticotomy Using Smartphone-Based Thermography: Reticulated Surgical Guide vs Dynamic Navigation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: URomLS_Thermography
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Orthodontic Tooth Movement; Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- static computer-guided surgery (Active Comparator)
  Interventions: Procedure: static computer-guided Corticotomy; Diagnostic Test: smartphone-based thermography
- dynamic computer guided-surgery (Experimental)
  Interventions: Procedure: dynamic computer-guided Corticotomy; Diagnostic Test: smartphone-based thermography

INTERVENTIONS:
Procedure: dynamic computer-guided Corticotomy — corticotomy cuts were made guided by a dynamic navigation system, ensuring accuracy and reducing the risk of injuries
  Arms: dynamic computer guided-surgery
Procedure: static computer-guided Corticotomy — corticotomy cuts were made guided by a static system (using reticulated surgical template), ensuring accuracy and reducing the risk of injuries
  Arms: static computer-guided surgery
Diagnostic Test: smartphone-based thermography — a Mini2 Infrared Smartphone Camera (Hangzhou HIKMICRO Sensing Technology Co., China) was initially calibrated with the surrounding ambient temperature. The calibration phase was essential as it enabled the device's algorithm to have a reference point based on the surrounding conditions and eliminate any bias caused by varying environmental temperatures. Then, pre-operative temperatures of attached gingiva and alveolar mucosa surfaces were recorded. The measurements were registered by distinguishing, for both arches, the temperature corresponding to soft tissues from incisor region (from central incisor to homolateral canine), premolar region (first and second premolars), and molar region (first and second molars).

SUMMARY:
Objectives:

The aim of the present split-mouth randomized clinical trial was to compare the effectiveness of two innovative corticotomy techniques, using reticulated static computer-guided surgery and dynamic computer-guided surgery, in terms of prevention of tissue overheating.

Material and Methods:

Four adult subjects requiring accelerated orthodontic treatment were enrolled. Each subject received both interventions in different quadrants. Preoperative surgical planning involved cone-beam computed tomography (CBCT) and optical scanning to superimpose DICOM and STL files. The static technique utilized a digitally designed reticulated surgical guide featuring multiple irrigation holes, while the dynamic technique employed a navigation system to provide real-time guidance. Preoperative, intraoperative and immediate postoperative tissue temperatures were recorded using an infrared smartphone camera. Statistical analyses, including Student's t-test, Mann-Whitney, and Welch tests, were performed to assess differences in thermographic measurements.

DETAILED DESCRIPTION:
The aim of the present study was to compare the effectiveness of two innovative corticotomy techniques, using reticulated static computer-guided surgery and dynamic computer-guided surgery, in terms of prevention of tissue overheating.

The initial hypothesis was that there were no statistically significant differences between the temperatures generated during the corticotomy between the two techniques used.

The present split-mouth randomized pilot clinical trial was conducted, in accordance with the ethical principles of the Declaration of Helsinki and CONSORT guidelines at the Department of Oral and Maxillofacial Sciences of Sapienza University of Rome, from October 2024 to February 2025. The patients were informed of the content, risks and benefits of the study, and written consent was obtained. The investigation received approval from the Ethics Committee of Lazio Area 1 (no. 7782).

The eligibility criteria were: (1) age >18 years, (2) need for orthodontic treatment and request of short-term orthodontic treatment, (3) good oral hygiene, (4) absence of systemic and oral cavity acute infection, (5) good general health.

The exclusion criteria were as it follows: (1) uncontrolled systemic disease; (2) syndromic patients; (3) smoking habit; (4) periodontal disease.

Based on the inclusion criteria, 4 patients were included and treated. The quadrant of the two corticotomy techniques was randomly decided by a coin toss and carried out by people unrelated to the research. The surgical procedure was performed by a single experienced operator (MC).

In order to achieve a shorter duration of orthodontic therapies and a safe and minimally invasive procedures, computer-assisted corticotomies were planned and performed using, in the same subject but in different quadrants, reticulated static computer-guided surgery and dynamic computer-guided surgery.

Each subject, after an intraoral examination and periodontal health assessment, underwent cone-beam computed tomography (CBCT) examination of the jaws and optical scanning. DICOM (Digital Imaging and COmmunications in Medicine) and STL (Standard Triangulation Language) files were superimposed to determine appropriate sites.

CBCT images were taken using the Scanora 3Dx cone-beam device (Soredex, Tuusul, Finland) and the exposure parameters were: 10 mA, 90 kV, 10 mA, total scanning time of 15.0 seconds, effective radiation time of 4.0 seconds, voxel size of 0.2 mm, field of view limited to upper and lower jaws. The STL files were collected using the Medit i700 intraoral scanner (Medit, Seoul, South Korea).

Once the superposition was performed, the corticotomy cuts were planned for each quadrant according to the randomly assigned technique. Regardless of the assigned technique, the space between the root of each tooth was assessed, and a longitudinal axis, running parallel to each root was established. Further, the surgical cuts were planned at a distance of at least 2 mm from the papilla, penetrating through the thickness of the cortical layer entirely. The cuts were designed on the basis of the use of the OT7A piezoelectric cutting insert (Mectron, Carasco, Genoa, Italy), considering a 0.75 mm dimension of the micro-saw.

The areas treated using static computer-guided technique involved the use of reticulated surgical guides -i.e. surgical guides characterized by slots to guide the piezoelectric saw and several holes to allow irrigation - designed through the use of Implant 3D software (Media Lab Spa, Milan, Italy). The 3D STL model of the reticulated surgical guide was printed using a Zortrax Inkspire 3D printer (Zortrax S.A. w restrukturyzacji, Olsztyn, Poland) and the Raydent surgical guide resin (Zortrax S.A. w restrukturyzacji, Olsztyn, Poland).

On the other hand, areas treated by dynamic computer-guided technique involved the use of the Navident dynamic navigation system (ClaroNav Technology Inc, Toronto, Canada).

The surgical phase began by asking the patient to rinse with 0.2% chlorhexidine mouthwash for 1 minute pre-operatively and then upper and lower plexus anesthesia was performed using mepivacaine with adrenaline 1:100.000 (Molteni Farmaceutici, Scandicci, Florence, Italy). Subsequently, in order to enable the use of the dynamic navigation system, two reference pattern tags - Head tracker and Jaw tracker - were temporarily fixed on the subject, and a calibration phase began selecting, for each jaw, three reference points on the 3D reconstruction of DICOM file generated by the Navident software (ClaroNav Technology Inc, Toronto, Canada). A calibration accuracy check was performed prior to the surgical phase, ensuring acceptable deviation values of ≤0.5 mm.

At this point, a Mini2 Infrared Smartphone Camera (Hangzhou HIKMICRO Sensing Technology Co., China) was initially calibrated with the surrounding ambient temperature. This calibration phase was essential as it enabled the device's algorithm to have a reference point based on the surrounding conditions and eliminate any bias caused by varying environmental temperatures. Then, pre-operative temperatures of attached gingiva and alveolar mucosa surfaces were recorded. The measurements were registered by distinguishing, for both arches, the temperature corresponding to soft tissues from incisor region (from central incisor to homolateral canine), premolar region (first and second premolars), and molar region (first and second molars).

After that, the reticulated surgical guides were positioned, and their stability was checked. Vertical gingival incisions were made interpromiximally below the interdental papilla in the two quadrants treated with static computer-guided surgery using a number 11 scalpel blade, and corticotomy cuts were performed using the Mectron Piezosurgery White (Mectron, Carasco, Genoa, Italy) piezoelectric surgical device and OT7A piezoelectric cutting insert (Mectron, Carasco, Genoa, Italy).

For the remaining quadrants, a vertical full-thickness gingival incision, below the interdental papilla, was performed using a number 11 scalpel blade by using the dynamic system. The OT7A micro-saw was calibrated and a calibration accuracy check was executed also in this phase, and thereafter, corticotomy cuts were performed following the real-time indications of the relative position of the micro-saw as indicated by the software, following the virtual planning made in the planning phase.

During the execution of the corticotomy cuts, for each technique used, the same flow and temperature of the cooling liquid was used, and intra-operative temperatures were recorded through the infrared smartphone camera. In addition, the post-operative tissue temperatures were registered also immediately after the corticotomies were performed.

Each thermographic measurement was performed by a single calibrated operator (A.P.) , at the same distance from subjects' soft tissues (30 centimeters) during the entire surgical time.

Statistical analysis was performed using Excel (Microsoft, Redmond, Washington, USA) and the statistical software package SPSS version 27.0 (IBM Corp., New York, USA).

To reduce the risk of statistical analysis bias, a blinded statistician external to the research performed the statistical analysis.

Results were described using descriptive statistics (including mean, minimum, maximum values and standard deviations).

The Shapiro-Wilk normality test and Brown-Forsythe test were used to assess the distribution of the data and the equality of variances, respectively. Violations of the normality or equal variance assumptions were detected for certain parameters.

The Student T-test was performed for variables without violation of assumptions, while Mann-Whitney test and Welch test were carried out, respectively, for non-normal distributed data and unequal variance variables.

The level of significance was set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* need for orthodontic treatment and request of short-term orthodontic treatment,
* good oral hygiene,
* absence of systemic and oral cavity acute infection,
* good general health.

Exclusion Criteria:

* uncontrolled systemic disease;
* syndromic patients;
* smoking habit;
* periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Quantitative Surface Temperature Assessment via Smartphone-Based Infrared Thermography. | From the start to the end of the surgical treatment
  The measurement, done using smartphone-based thermal camera, involves capturing standardized baseline and follow-up thermal images of defined body regions (in this case attached gingiva and oral mucosa), with temperature values recorded as the mean of three consecutive readings. The data will be further aggregated using mean and standard deviation metrics for comparative analysis over time and between study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Sciences Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No